CLINICAL TRIAL: NCT00253409
Title: Mesothelioma and Radical Surgery Trial
Brief Title: Combination Chemotherapy With or Without Surgery and Radiation Therapy in Treating Patients With Mesothelioma That Can Be Removed By Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000448615; ICR-CTSU-MARS; EU-20532
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Drug Therapy; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: chemotherapy
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy before surgery may shrink the tumor so that it can be removed. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether combination chemotherapy is more effective with or without surgery and radiation therapy in treating mesothelioma.

PURPOSE: This randomized clinical trial is studying combination chemotherapy, surgery, and radiation therapy to see how well they work compared to combination chemotherapy alone in treating patients with mesothelioma that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the feasibility of neoadjuvant combination chemotherapy with vs without surgery and adjuvant radiotherapy in patients with resectable malignant mesothelioma.
* Compare the overall survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a multicenter, pilot study followed by a randomized, controlled study.

Patients undergo 3 courses of a platinum-based (cisplatin or carboplatin) combination chemotherapy regimen to be determined by the treatment center. Upon completion of combination chemotherapy, patients are randomized to 1 of 2 treatment arms provided tumor is resectable and there is no disease progression.

* Arm I: Patients undergo extra-pleural pneumonectomy followed by post-operative radiotherapy.
* Arm II: Patients undergo follow-up only. Patients may receive additional standard therapy according to their treatment center.

Quality of life is assessed at baseline, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

After completion of study treatment, patients are followed periodically for 2 years and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 50-670 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and immuno-histochemically confirmed malignant mesothelioma

  * Resectable disease (T1-3, N0-1, M0) with no distant metastases
* Eligible to undergo extra-pleural pneumonectomy based on British Thoracic Society guidelines

PATIENT CHARACTERISTICS:

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Normal renal function

Cardiovascular

* Ejection fraction ≥ 40%

Pulmonary

* Predicted post-operative FEV_1 ≥ 40%
* Predicted post-operative DLCO ≥ 40%
* No significant pulmonary hypertension

Other

* No physical or personal condition that would preclude ability to undergo chemotherapy or post-operative radiotherapy
* No physical or personal condition that would preclude ability to comply with follow-up requirements

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2005-05; Primary Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Peckitt, Study Chair — Institute of Cancer Research, United Kingdom
Locations (17):
- United Kingdom (17):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Bristol Royal Infirmary, Bristol, England
  - Queen's Hospital, Burton-on-Trent, England
  - Addenbrooke's Hospital, Cambridge, England
  - Papworth Hospital, Cambridge, England
  - Ipswich Hospital, Ipswich, England
  - Cookridge Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Glenfield Hospital, Leicester, England
  - St. Thomas' Hospital, London, England
  - Royal Marsden - London, London, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Institute of Cancer Research - Sutton, Sutton, England
  - Royal Marsden - Surrey, Sutton, England